CLINICAL TRIAL: NCT03829774
Title: To Study and Evaluate the Effectiveness of Treatment by Percutaneous Electrical NeuroStimulation (PENS) for Post-operative Pain in Cesarean Section Patients Using Primary Relief v 2.0
Acronym: POPS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: DyAnsys, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CS/PRv2.0/C-Sec/2019
Record Dates: First submitted 2019-01-27; First posted 2019-02-04 (Actual); Last update posted 2019-02-05 (Actual); Status verified 2019-01

CONDITIONS: Cesarean Section; Dehiscence
MeSH Terms: interventions — Acetaminophen

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Primary Relief v 2.0 Device (Experimental): The test product or device called Primary Relief v 2.0 device will be used for the study. The study will be conducted for a period of two to three months with the treatment period of 3 - 4 days i.e single treatment (installation). The additional time taken will be to define the characteristics of the patient population and to recruit appropriate patients. Finally, there will be a data analysis and report writing period. Overall, the study is expected to 3 months. The device will be placed onto the auricle part of the ear for percutaneous electrical nerve stimulation.
  Interventions: Device: Primary Relief v 2.0
- Paracetamol (Placebo Comparator): A control group, receiving a standard treatment as follows: primary choice of analgesic was intravenous Paracetamol , 1 gram, and if the pain relief was inadequate, diclofenac inj. If pain persisted in spite of these measures, 50 mg tramadol was administered intravenously
  Interventions: Drug: Paracetamol

INTERVENTIONS:
Device: Primary Relief v 2.0 — The test product or device called Primary Relief v 2.0 will be used for the study. The study will be conducted for a period of two to three months with the treatment period of 3 - 4 days i.e single treatment (installation). The additional time taken will be to define the characteristics of the patient population and to recruit appropriate patients. Finally, there will be a data analysis and report writing period. Overall, the study is expected to 3 months. The device will be placed onto the auricle part of the ear for percutaneous electrical nerve stimulation.
  Other Names: Percutaeneous Nerve Field Stimulator Neurostimulator
  Arms: Primary Relief v 2.0 Device
Drug: Paracetamol — A control group, receiving a standard treatment as follows: primary choice of analgesic was intravenous paracetamol, 1 gram, and if the pain relief was inadequate, diclofenac inj. If pain persisted in spite of these measures, 50 mg tramadol was administered intravenously
  Other Names: Standard Drug Treatment for Postoperative pain
  Arms: Paracetamol

SUMMARY:
To study and evaluate the Effectiveness of Treatment by Percutaneous Electrical NeuroStimulation (PENS) for post-operative pain in Cesarean Section patients using First Relief

ELIGIBILITY:
Inclusion Criteria:

1. Age range between 22 - 35 years
2. Patient willing to undergo C-section surgery
3. Patient having pains after one hour of post C-Section surgery
4. Patients who is conscious and oriented for device installation after anesthetic effect
5. Patient who completed required clinical and biochemical investigations as deemed necessary by the gynecologist after post C - section surgery.
6. No previous poor obstetrical outcome
7. No experience in Han's Acupoint nerve stimulator and TENS for other reasons.
8. Term pregnancy (> 37 weeks of gestation).
9. Understands and is willing to participate in the clinical study and can comply with study procedures.
10. Normal cognitive and communicative ability as judged by clinical assessment and ability to complete self-reported questionnaires.

Exclusion Criteria:

1. Had been diagnosed with other diseases such as preoperative presence of maternal mental, neurological disease, affecting evaluation of pains and disease condition.
2. Had combined with gestational hypertension, gestational diabetes, gestational thyroid disease.
3. Had taken analgesic drugs
4. Had used diazepam, piperazine hydrochloride or other sedative, analgesic drugs in the stage of labor.
5. Were overweight or low pregnancy weight, Body mass index (< 18.5 or >25 kg/m2).
6. Patients who are not agreeing to receive painless labor and not sign the informed consent form.
7. Neonatal problem requiring immediate separation from the mother for medical care or NICU admittance.
8. Severe placental abruption.
9. Hydrops (accumulation of fluid or edema in fetus body tissue and cavities) if secondary to anemia or heart failure.
10. Known twin to twin transfusion syndrome (TTS).
11. Congenital anomalies that may hamper the procedure (gastroschisis, amphalacele, spina bifida).
12. Home birth.
13. Severe mental health problem
14. Hearing impairment.
15. Legal abortion
16. Twin pregnancy
17. Instrumental birth
18. Uterine anomalies with contraindication for vaginal birth. Eg: previous opening of uterine cavity, myomectomy, congenital abnormalities.
19. Placenta anomalies.
20. Placenta praevia, suspected acreta, increta, percreta especially after previous caesarean.
21. Fetal abnormalities, growth restriction.
22. Maternal complication with surgery.
23. Subjects on any investigational drug(s) or therapeutic device(s) within 30 days preceding screening; or subject or physician anticipates use of any of these therapies by the subject during the course of the study
24. Previous participation in the Treatment Phase of this Protocol
25. Malignant disease not in remission for five years or more that has been medically or surgically treated without evidence of metastases
26. Presence of one or more medical conditions, as determined by medical history, which seriously compromises the subject's ability to complete the study, including history of poor adherence with medical treatment, unstable pain intensity or pain medications 6 weeks prior to the study, renal, hepatic, hematologic, active auto-immune or immune diseases that, in the opinion of the Investigator, would make the subject an inappropriate candidate for this study: a) One or more abnormal blood biochemistry analyte result that is ≥ 3 times that of the upper limit of the normal range
27. Known history of having Acquired Immunodeficiency Syndrome (AIDS) or with a history known to be infected with Human Immunodeficiency Virus (HIV)
28. American Heart Association (AHA) Class III and IV congestive heart failure (CHF), as defined by the following criteria: a) Class III: Symptoms with moderate exertion b) Class IV: Symptoms at rest or c) Cardiac pacemakers.
29. Subjects with a diagnosis of psychiatric disorders such as major depressive disorder, bipolar disorder, obsessive compulsive disorder, generalized anxiety, dysthymia or suicidality/suicide ideation
30. Subjects not willing to undergo treatment before discharge from the hospital.

Ages: 22 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Pregnant Women willing to undergo C-Section
Enrollment: 22 (Estimated)
Dates: Start 2019-01-02 (Actual); Primary Completion 2019-03 (Estimated); Study Completion 2019-07 (Estimated)

PRIMARY OUTCOMES:
assessing the effects of PENS therapy in Postoperative period of Lower Segment Caesarean Section pain using VAS score. | 2 hours of device activation
  To assess the effects of PENS therapy in Post-Operative period of Lower Segment Caesarean Section pain using the Visual Analogue Scale measurement. The level of pain is calculated from the VAS (Visual Analogue Scale) before the device is installed and assessed after 2 hours of the device activation. The pain level should be decreased when assessing after 2 hours of device installation. The score should be below 5. where 0 being no pain, 5 being moderate and 10 being maximum pain.

SECONDARY OUTCOMES:
Evaluate the impact of this treatment in terms of Quality Of Life | 2nd day
  whether treatment can negate the need for more complex surgical treatments and/or reduce the need for drug treatment. Change in quality of life will be measured using the Evaluation form measurement.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinic, Warangal, Telangana, India

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Zimpel SA, Torloni MR, Porfirio GJ, Flumignan RL, da Silva EM. Complementary and alternative therapies for post-caesarean pain. Cochrane Database Syst Rev. 2020 Sep 1;9(9):CD011216. doi: 10.1002/14651858.CD011216.pub2. PMID 32871021